CLINICAL TRIAL: NCT04506372
Title: Angiotensin-converting Enzyme Inhibitors and Angiotensin Receptor Blockers During the Perioperative Period: to Withdraw or to Continue? A Multicenter Randomized Controlled Trial
Brief Title: Management of Angiotensin Inhibitors During the Perioperative Period
Acronym: AIPOP
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: slow recruitment rate
Sponsor: UMC Utrecht (Other)
Collaborators: ZonMw: The Netherlands Organisation for Health Research and Development (Other)
Responsible Party: Principal Investigator, Judith van Waes, J.A.R. van Waes, MD PhD, UMC Utrecht
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: AIPOP
Record Dates: First submitted 2020-08-06; First posted 2020-08-10 (Actual); Last update posted 2023-11-29 (Actual); Status verified 2023-11

CONDITIONS: Surgery; Angiotensin Hypertension; Perioperative Complication
Keywords: Noncardiac surgery; Angiotensin inhibitors; Perioperative management
MeSH Terms: interventions — Blood Specimen Collection

STUDY DESIGN:
Intervention Model Description: Randomized controlled clinical trial
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): Perioperative withdrawal of ACEI/ARB.
  Interventions: Drug: Perioperative withdrawal of angiotensin converting enzyme inhibitors and angiotenin receptor blockers; Diagnostic Test: Blood draw; Behavioral: Diary to register drug adherence; Behavioral: Quality of life questionnaire; Behavioral: WHODAS questionnaire
- Control group (Active Comparator): Perioperative continuation of ACEI/ARB.
  Interventions: Diagnostic Test: Blood draw; Behavioral: Diary to register drug adherence; Behavioral: Quality of life questionnaire; Behavioral: WHODAS questionnaire

INTERVENTIONS:
Drug: Perioperative withdrawal of angiotensin converting enzyme inhibitors and angiotenin receptor blockers — Withdrawal from 24 hours before surgery until 24-48 hours after surgery. The ACEI/ARB medication is resumed on the second or third day after surgery, as soon as the clinical condition allows based on judgement by the attending physician.
  Arms: Intervention group
Diagnostic Test: Blood draw — Blood will be drawn to measure creatinin and troponin: once before surgery, on the first and second postoperative day, and within 4-8 weeks after surgery
Behavioral: Diary to register drug adherence — To register medication adherence, patients will be asked to fill out their medication intake (of ACEI/ARB) in a diary from a week before surgery until surgery.
Behavioral: Quality of life questionnaire — Patients are asked to fill out a quality of life questionnaire (EQ-5D) before surgery and at three months after surgery
Behavioral: WHODAS questionnaire — Patients are asked to fill out a questionnaire about disabilities (WHO Disability Assessment Schedule 2.0) before surgery and at three months after surgery

SUMMARY:
This is a multicenter randomized clinical trial to determine the effect of continuation versus withdrawal of angiotensin-converting enzyme inhibitors (ACEI) and angiotensin receptor blockers (ARB) in the perioperative period on postoperative complications.

DETAILED DESCRIPTION:
Rationale:

Angiotensin inhibitors including angiotensin convertying enzyme inhibitors (ACEI), and angiontensin receptors blockers (ARB) are frequently used to treat patients with chronic hypertension. These drugs reduce morbidity and mortality on the long term. However, when patients who use ACEI or ARB undergo surgery, hypotension may occur in the perioperative period, which may can lead to organ hypoperfusion and damage. On the other hand, when ACEI and ARB are temporarily discontinued in the perioperative period, hypertension may occur which also may lead to complications. Therefore, before surgery the anesthesiologist advises the patient to continue or to temporarily withdraw this drug. Importantly, it is currently unclear which strategy is best, and international guidelines are disconcordant on this point. Policy varies between hospitals and even between anesthesiologists: in some hospitals, patients are advised to temporarily withdraw the ACEI/ARB, whilst in other hospitals patients are advised to continue this drug. The latest research on this topic suggests that perioperative continuation of ACEI/ARB may lead to more complications, but definitive evidence is lacking. Therefore it is important to perform a randomized trial to compare the two options: perioperative continuation versus withdrawal of ACEI/ARB.

Objective:

The objective of this trial is to determine the effect of continuation versus withdrawal of ACEI and ARB in the perioperative period on postoperative complications, expressed as acute kidney injury (AKI), myocardial injury, and quality of life (QoL).

Study design:

This is a multicenter randomized clinical trial.

Study population:

Patients who use ACEI/ARB chronically for treatment of hypertension and who are scheduled for an elective intermediate to high risk non-cardiac surgical procedure with an expected postoperative length of hospital stay of at least 2 days, are eligible for inclusion. Patients who use a combination pill of ACEI/ARB with a diuretic are eligible as well. Patients who use a combination pill ACEIwith another drug will be excluded, as well as patients who use other drugs acting on the renin aldosterone angiotensin system.

Intervention:

The intervention is the withdrawal of ACEI/ARB in the perioperative period, i.e. 24 hours before surgery until 24-48 hours after surgery. The ACEI/ARB medication is resumed on the second or third day after surgery, as soon as the clinical condition allows based on judgement by the attending physician.

This intervention will be compared to perioperative continuation of ACEI/ARB.

Main study parameters/endpoints:

The primary outcome for this study is postoperative acute kidney injury, defined according to the Kidney Disease Improving Global Outcomes (KDIGO) guideline.

Secondary outcomes include postoperative myocardial injury, intraoperative and postoperative hypotension and hypertension, length of stay in the hospital or nursing home, kidney function loss and end-stage renal disease within three months after surgery, major cardiovascular complications (myocardial infarction, coronary revascularization, heart failure, arrhythmia, stroke) within three months after surgery, all-cause mortality within three months after surgery and a quality of life (QoL) assessment.

ELIGIBILITY:
Inclusion Criteria:

* Chronic ACEI or ARB use for the treatment of hypertension. Patients who use a com-bination pill with a diuretic are eligible as well;
* Scheduled for elective intermediate to high risk noncardiac surgery, defined according to the European Society of Cardiology / European Society of Anesthesiology guidelines on noncardiac surgery;
* Expected postoperative length of stay of at least two days.

Exclusion Criteria:

* Severe chronic kidney disease, defined as GFR<30 ml/min/1.73 m2;
* ACEI/ARB use for the treatment of chronic systolic heart failure, defined as left ven-tricular ejection fraction ≤40%;
* ACEI/ARB use within one year after ST-elevated myocardial infarction, according to the fourth universal definition of myocardial infarction;
* Transplant surgery;
* ACEI/ARB use in a combination pill together with a drug other than a diuretic, including calcium channel blockers, beta-blockers and neprilysin inhibitors;
* Use of drugs acting on the renin-angiotensin-aldosterone system other than ACEI/ARB, e.g. aliskiren.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 342 (Actual)
Dates: Start 2020-09-11 (Actual); Primary Completion 2023-02-06 (Actual); Study Completion 2023-09-01 (Actual)

PRIMARY OUTCOMES:
Postoperative acute kidney injury | Within two days after surgery
  Postoperative acute kidney injury, defined according to the Kidney Disease Improving Global Outcomes (KDIGO) guideline.

SECONDARY OUTCOMES:
Postoperative myocardial injury | Within two days after surgery
  Postoperative myocardial injury, defined as an increased level of serum troponin above the clinical cut-off value
Acute postoperative myocardial injury | Within two days after surgery
  Acute postoperative myocardial injury, defined as an absolute postoperative increase in serum troponin of more than clinical cut-off value as compared to the preoperative value
Intraoperative hypotension | From the start of anesthesia until the end of surgery
  Intraoperative hypotension, defined as a mean arterial pressure <65 mmHg for at least 10 minutes
Postoperative hypotension | From the end of surgery up to and including the second postoperative day
  Postoperative hypotension, defined as a mean arterial pressure <65 mmHg
Preoperative hypertension | Within 24 hours before start of anesthesia
  Preoperative severe hypertension, defined as blood pressure >180/110 mmHg
Postoperative hypertension | From the end of surgery up to and including the second postoperative day
  Postoperative severe hypertension, defined as blood pressure >180/110 mmHg
Length of stay | Within three months after surgery
  Length of stay in hospital or nursing home
Kidney function loss | Within three months after surgery
  Decline in glomerular filtration rate as compared to before surgery
Acute kidney function loss | Within two days after surgery
  Decline in glomerular filtration rate as compared to before surgery
End-stage renal disease | Within three months after surgery
  End-stage renal disease, defined as renal disease requiring dialysis or organ transplantation
Major cardiovascular complications | Within three months after surgery
  Major cardiovascular complications (myocardial infarction, coronary revascularization, heart failure, arrhythmia, stroke)
Mortality | Within three months after surgery
  All-cause mortality
Quality of life | At three months after surgery
  Quality of life based on the EuroQoL 5D questionnaire
Disability | At three months after surgery
  Disability at three months after surgery based on the World Health Organization Disability Activity Score (WHODAS):
  * Change in WHODAS as compared to before surgery (continuous measure);
  * Clinically important change in WHODAS defined as an increase of 5% or more as compared to before surgery;
  * Disability free survival defined as WHODAS <16%;
  * Clinically important disability defined as WHODAS >35%.

CONTACTS AND LOCATIONS:
Overall Officials: Judith van Waes, MD PhD, Principal Investigator — UMC Utrecht; Wilton van Klei, MD PhD, Principal Investigator — UMC Utrecht
Locations (7):
- University Health Network Toronto, Toronto, Ontorio, Canada
- Netherlands (6):
  - Amsterdam UMC location AMC, Amsterdam
  - Amsterdam UMC location VU, Amsterdam
  - Amphia Hospital, Breda
  - Antonius Hospital, Nieuwegein
  - Erasmus MC, Rotterdam
  - UMC Utrecht, Utrecht

REFERENCES:
- See also: Related Info — https://www.umcutrecht.nl/en/ziekenhuis/wetenschappelijk-onderzoek/aipop-management-of-angiotensin-inhibitors-during-the-perioperative-period